CLINICAL TRIAL: NCT04905212
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study of Telitacicept for Injection (RC18) With an Optional Open Label Extension in Subjects With IgA Nephropathy
Brief Title: A Study of Telitacicept for Injection (RC18) in Subjects With IgA Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision that continuing with the study would not generate useful data
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC18G004
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: IgA Nephropathy
Keywords: Berger Disease; Berger's Disease; IGA Glomerulonephritis; IGA Nephropathy; Primary IGA Nephropathy; Immunoglobulin A Nephropathy Nephritis; IGA Type Nephropathy, IGA
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Telitacicept 160mg (Experimental): Telitacicept 160mg subcutaneous injection once weekly, and a total of 24 doses
  Interventions: Drug: Telitacicept 160mg
- Telitacicept 240mg (Experimental): Telitacicept 240mg subcutaneous injection once weekly, and a total of 24 doses
  Interventions: Drug: Telitacicept 240mg
- Placebo (Placebo Comparator): Placebo subcutaneous injection once weekly, and a total of 24 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telitacicept 160mg — Subcutaneous injection Telitacicept 160mg. The injection site can be at the thigh, abdomen, or upper arm.
  Arms: Telitacicept 160mg
Drug: Telitacicept 240mg — Subcutaneous injection Telitacicept 240mg. The injection site can be at the thigh, abdomen, or upper arm.
  Arms: Telitacicept 240mg
Drug: Placebo — Subcutaneous injection placebo. The injection site can be at the thigh, abdomen, or upper arm.
  Arms: Placebo

SUMMARY:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled clinical study with an optional open label extension to evaluate the safety and efficacy of Telitacicept for Injection (RC18) in the treatment of IgA nephropathy.

DETAILED DESCRIPTION:
IgA nephropathy is a kidney disease in which IgA, a protein meant to defend the body against foreign invaders, accumulates in the kidneys and damages them. This study will seek to determine the safety and efficacy of Telitacicept for Injection (RC18) in the treatment of IgA nephropathy.

The study is composed of 4 parts: a screening period, a double-blind treatment period, an optional open label extension, and a follow-up period. Subjects with confirmed IgA nephropathy will be enrolled and randomized 1:1:1 to Telitacicept 160 mg, Telitacicept 240 mg, or placebo (10 per arm).

ELIGIBILITY:
Inclusion Criteria:

1. IgA nephropathy confirmed by pathological biopsy;
2. Male or female aged ≥ 18 years old;
3. Average 24-hour urine total protein ≥ 0.75 g/24 h
4. Estimated GFR (using the CKD-EPI formula) > 30 mL/min per 1.73 m^2;
5. Stabilized AEI/ARB medications, diuretics, or other antihypertensive therapy.

Exclusion Criteria:

1. Patients with clinically significant abnormal laboratory tests at screening;
2. Evidence of rapid eGFR decrease > 15 ml/min during screening;
3. Renal or other organ transplantation prior to, or expected during, the study;
4. Patients with secondary IgA nephropathy;
5. Patients with nephrotic syndrome, crescentic nephritis minimal change nephropathy with IgA deposition, or other pathological or clinical types of renal diseases that may confound the study data interpretation;
6. Patients with history of any severe unstable cardiovascular and cerebrovascular events within 12 weeks prior to screening;
7. Immunocompromised individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24-hour urine protein at Week 24. | Week 24
  Change from baseline in urine protein over 24 hours to Week 24 will be measured

SECONDARY OUTCOMES:
Change from baseline in estimated glomerular filtration rate (eGFR) at Weeks 4, 8, 12, 16, 20, 24, 32, 36 and 48 | Weeks 4, 8, 12, 16, 20, 24, 32, 36 and 48
  Change from baseline in eGFR by visit
Change from baseline in urine protein-to-creatinine ratio (UPCR) and urine albumin-to-creatinine ratio (UACR) at Weeks 4, 8, 12, 16, 20, 24, 32, 36, and 48; | Weeks 4, 8, 12, 16, 20, 24, 32, 36, and 48
  Change from baseline in Urine protein-to-creatinine ratio (UPCR) and Urine albumin-to-creatinine ratio (UACR) by visit.
Change from baseline in immunological parameters (IgA, IgG, IgM, C3, C4, and B lymphocytes) at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 48, and EOT visit. | Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 48, and EOT visit.
  Changes from baseline in Immunoglobulins (IgA, IgG, IgM), B lymphocytes (CD19+), complements (C3, C4)

OTHER OUTCOMES:
The incidence and severity of adverse events | 27 weeks
  Number and intensity of adverse events
Immunogenicity endpoints | Week 0, 4, 8, 12, 16, 20, 24 and 27
  Anti-drug antibody (ADA), incidence, titers and duration
Biomaker endpoints serum concentration | Week 0, 4, 8, 12, 16, 20, and 24
  BLyS serum concentration, APRIL serum concentration, and BLyS-drug complex
Pharmacokinetic endpoints | Week 0, 4, 8, 12, 16, 20, 24 and 27
  Free Telitacicept serum concentration and total Telitacicept serum concentration

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Remegen Site #5, Los Angeles, California
  - Remegen Site #13, Los Angeles, California
  - Remegen Site #14, Los Angeles, California
  - Remegen Site #10, Sacramento, California
  - Remegen Site #8, San Francisco, California
  - Remegen Site #16, Fort Lauderdale, Florida
  - Remegen Site #17, Augusta, Georgia
  - Remegen Site #2, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639